CLINICAL TRIAL: NCT00097890
Title: An Open Label Six-Month Maintenance Clinical Trial of Replagal Enzyme Replacement Therapy in Patients With Fabry Disease Who Have Completed TKT027
Brief Title: Replagal Enzyme Replacement Therapy for Adults With Fabry Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050046; 05-N-0046
Record Dates: First submitted 2004-11-30; First posted 2004-12-01 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-12

CONDITIONS: Fabry Disease
Keywords: Lysosomes; Storage; Glycolipid; Fabry Disease; Stroke
MeSH Terms: conditions — Fabry Disease; Stroke | interventions — agalsidase alfa

INTERVENTIONS:
Drug: Replagal (Agalsidase Alfa)
Drug: Replagal

SUMMARY:
This study will determine the safety and effectiveness of the drug Replagal for treating people with Fabry disease, an inherited metabolic disorder. In this disease, an enzyme called alpha-galactosidase A, which normally breaks down a lipid (fatty substance) known as ceramidetrihexoside, is missing or does not function properly. As a result, the lipid accumulates in the body, causing problems with the kidneys, heart, nerves, and blood vessels. This study will examine whether replacing the missing alpha-galactosidase A with a genetically engineered form of the enzyme called Replagal can reverse the illness.

Patients with Fabry disease who are 18 years of age or older and have completed 10 weeks of Replagal therapy as participants in protocol TKT027 may be eligible for this 6-month study extension.

Participants undergo the following tests and procedures:

* Intravenous (IV) infusions of Replagal every other week over 25 weeks for a total of 13 infusions, with close monitoring during and after the infusions.
* Brief safety evaluations at the time of each infusion, including a check of vital signs (blood pressure, pulse, breathing rate, temperature), review of any side effects, and review of medications.
* Comprehensive evaluations at baseline (before starting Replagal therapy), after 13 and 25 weeks of therapy, and 30 days after completing therapy. These include a medical history and physical examination, symptoms and pain questionnaire, blood and urine tests, check of vital signs, electrocardiogram (EKG), 2-hour Holter monitor, and sweat test (QSART).

DETAILED DESCRIPTION:
Objectives: To evaluate the safety of the current standard Replagal treatment regimen of 0.2 mg/kg given intravenously every two weeks over an additional 6 months in patients who have completed 10 weeks of Replagal therapy in the TKT027 study.

Study Population: Hemizygous males with Fabry disease who are 18 years of age or older who have completed 10 weeks of Replagal therapy in TKT027.

Design: This is an open-label, multi-center study that will assess the safety of 0.2 mg/kg every two weeks of enzyme replacement therapy with Replagal.

ELIGIBILITY:
INCLUSION CRITERIA:

Subject must have completed 10 weeks of infusions in Study TKT027 with intent to complete participation in the study.

Subject must have adequate general health (as determined by the investigators) to undergo the specified phlebotomy regimen and protocol related procedures.

Subject must consent to participate in the protocol and must have voluntarily signed an Institutional Review Board/Independent Ethics Committee (IRB/IEC) approved informed consent form after all relevant aspects of the study have been explained and discussed with the patient.

EXCLUSION CRITERIA:

Subject is unable to understand the nature, scope, and possible consequences of the study.

Subject is unable to comply with the protocol, e.g., uncooperative with protocol schedule, refusal to agree to all of the study procedures, inability to return for safety evaluations, or is otherwise unlikely to complete the study, as determined by the investigator or the medical monitor.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25
Dates: Start 2004-11; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Brady RO, Gal AE, Bradley RM, Martensson E, Warshaw AL, Laster L. Enzymatic defect in Fabry's disease. Ceramidetrihexosidase deficiency. N Engl J Med. 1967 May 25;276(21):1163-7. doi: 10.1056/NEJM196705252762101. No abstract available. PMID 6023233
- [Background] Brady RO, Schiffmann R. Clinical features of and recent advances in therapy for Fabry disease. JAMA. 2000 Dec 6;284(21):2771-5. doi: 10.1001/jama.284.21.2771. PMID 11105184
- [Background] Meikle PJ, Hopwood JJ, Clague AE, Carey WF. Prevalence of lysosomal storage disorders. JAMA. 1999 Jan 20;281(3):249-54. doi: 10.1001/jama.281.3.249. PMID 9918480